CLINICAL TRIAL: NCT03778723
Title: Cerebral Oxygenation and Metabolism in Patients Undergoing Clipping of Cerebral Aneurysm: A Comparative Study Between Propofol-based Total Intravenous Anesthesia and Sevoflurane-based Inhalational Anesthesia
Brief Title: Effect of Propofol Midazolam on Cerebral Oxygenation and Metabolism During Clipping of Ruptured Cerebral Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD ∕17.08.07
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Ruptured Cerebral Aneurysm
MeSH Terms: interventions — Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia (TIVA) (Experimental): Patients will receive total intravenous anesthesia using Propofol and Midazolam
  Interventions: Drug: Total intravenous anesthesia (TIVA); Drug: Rescue fentanyl
- Inhalation Anesthesia (Active Comparator): Patients will receive Inhalation anesthesia using Sevoflurane
  Interventions: Drug: Inhalation Anesthesia; Drug: Rescue fentanyl

INTERVENTIONS:
Drug: Total intravenous anesthesia (TIVA) — Propofol (1.5-2 mg/kg/h) infusion, Midazolam (0.12 mg/kg/h) infusion
  Arms: Total intravenous anesthesia (TIVA)
Drug: Inhalation Anesthesia — Sevoflurane at a concentration of 2-2.5%
  Arms: Inhalation Anesthesia
Drug: Rescue fentanyl — Fentanyl in repeated doses (50 µg) when needed (heart rate or mean arterial blood pressure increase more than 20% of the basal value) are used for maintenance of analgesia

SUMMARY:
Despite the theoretical benefits of i.v. agents, volatile agents remain popular. In a study comparing desflurane, isoflurane, and sevoflurane in a porcine model of intracranial hypertension, at equipotent doses and normocapnia, cerebral blood flow (CBF) and ICP were least with sevoflurane.

Propofol is the most commonly used intravenous anesthetic. It has many theoretical advantages by reducing cerebral blood volume (CBV) and ICP and preserving both autoregulation and vascular reactivity. Neurosurgical patients anaesthetized with propofol were found to have lower ICP and higher CPP than those anaesthetized with isoflurane or sevoflurane.

The well known pharmacodynamic advantages of intravenous anesthetics may give this group of drugs superior cerebral effects when compared with inhalation anesthetics.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the cerebral hemodynamics and global cerebral oxygenation as well as the systemic hemodynamic changes using midazolam and propofol as total intravenous anesthetics (TIVA) in comparison with sevoflurane anesthesia in clipping of ruptured cerebral aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status III or IV.

Exclusion Criteria:

* Morbid obese patients.
* Severe or uncompensated cardiovascular diseases
* Severe or decompensated renal diseases
* Severe or decompensated hepatic diseases
* Severe or decompensated endocrinal diseases.
* Pregnancy
* Postpartum
* Lactating females
* Allergy to one of the agents used.
* Severely altered consciousness level.
* Sitting or prone position during surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Arterio-Jugular oxygen content difference | Immediately before and every 30 min for 6 hour following start of surgery
  The differences between arterial and jugular bulb oxygen contents
Estimated cerebral metabolic rate for O2 (eCMRO2) | Immediately before and every 30 min for 6 hour following start of surgery
  eCMRO2=Ca- jO2 x(PaCO2 ∕ 100), Where Ca jO2 is arterio-jugular O2 content difference. PaCO2 is arterial CO2 tension
Cerebral Extraction Rate of O2 (CEO2) | Immediately before and every 30 min for 6 hour following start of surgery
  Calculated as the differences between arterial and jugular bulb O2 saturations, CEO2 = SaO2 - SjvO2
Cerebral Blood Flow equivalent (CBFe) | Immediately before and every 30 min for 6 hour following start of surgery
  : Which is an index of flow metabolism relationship, calculated as a reciprocal of arterio-jugular O2 content difference. CBFe = 1 ∕CaO2-CjvO.

SECONDARY OUTCOMES:
Heart rate | Immediately before and every 30 min for 6 hour following start of surgery
Mean arterial blood pressure | Immediately before and every 30 min for 6 hour following start of surgery
Peripheral oxygen saturation | Immediately before and every 30 min for 6 hour following start of surgery
Central venous pressure | Immediately before and every 30 min for 6 hour following start of surgery
End tidal carbon dioxide tension | Immediately before and every 30 min for 6 hour following start of surgery
Sedation score | For 6 hours from induction of anesthesia
  - Postoperative level of sedation of all patients will be evaluated using Ramsay sedation scale
Time for first analgesic request from extubation | For 6 hours from induction of anesthesia
  Time for first analgesic request from extubation
Duration of stay in intensive care unit | For 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Mousa, MD, Study Chair — Professor; Mohammed A Ghanem, MD, Study Director — Associate Professor
Locations (1):
- Sherif A Mousa, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided